CLINICAL TRIAL: NCT01303471
Title: Pain Assessment During General Anesthesia : DOLANS (DOULeur ANeSthesie) Study
Brief Title: Pain Assessment During General Anesthesia
Acronym: DOLANS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 1008032; 2010-019591-67 (EudraCT Number)
Record Dates: First submitted 2011-02-18; First posted 2011-02-24 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-05

CONDITIONS: Pain
Keywords: pain assessment; anesthesia; analgesia; opioid; HRV; APV; autonomic nervous system (ANS); pupil size
MeSH Terms: conditions — Pain; Agnosia | interventions — Analgesics, Opioid; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- opioïd (Experimental): Different levels of remifentanyl of each group during nociceptive stimulation
  Interventions: Drug: opioid (remifentanyl)

INTERVENTIONS:
Drug: opioid (remifentanyl) — Infusion of remifentanyl (opioid) will be started at different levels for each group of the randomized study : 0 ng/ml (group 0), 1 ng/ml (group 1), 3 ng/ml (group 3) or 4 ng/ml (group 4)

SUMMARY:
During general anesthesia, two treatments are used : hypnotic and opioid treatment. Opioid treatment is used for pain assessment.

The change in haemodynamic variables and clinical sign are evaluated during anesthesia for pain assessment but these changes are not specific every time.

The main of this study is to investigate the relationship between calculated compartment concentration of remifentanil (opioid) and the parameters from HRV (Heart Rate Variability) and APV (Arterial Pressure Variability) before a standard noxious stimulation during general anesthesia at calibrated hypnosis level.

Our hypothesis is that nociceptive stimulation would have reproductible effects on HRV, and that these effects would be blunted or abolished by by adequate analgesia. The current study is thus designed to analyse HRV and APV in patients with stable hypnosis, before and during nociceptive surgical stimulation, at different levels of analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients under 55 years-old
* ASA status 1 or 2
* scheduled to undergo general anesthesia for different types of surgery (neurosurgical or medullar surgery, ear, nose or throat surgery or orthopedic surgery)

Exclusion Criteria:

* history of cardiac or autonomic disease
* diabetes
* obesity (BMI>30 kg/m2)
* medication altering autonomic nervous system tone
* history of eyes surgery

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2011-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HRV measurements during noxious stimulation | baseline and 5 minutes
  Analyse of HRV is a widely used, non-invasive technique to assess autonomic nervous system (ANS) activity. The typical spectral pattern of HRV includes two main spectral peaks : a low-freqency (LF) region, affected by both sympathetic and parasympathic activity, and a high-frequency (HF) peak centered at the respiratory frequency, which is associated with parasympathetic activity.
change from baseline in APV measurements during noxious stimulation | baseline and 5 minutes
  Analyse of APV is a widely used, non-invasive technique to assess autonomic nervous system (ANS) activity. The typical spectral pattern of APV includes two main spectral peaks : a low-freqency (LF) region, affected by both sympathetic and parasympathic activity, and a high-frequency (HF) peak centered at the arterial pressure, which is associated with parasympathetic activity.

SECONDARY OUTCOMES:
Change from baseline in pupil change during noxious stimulation | baseline and 5 minutes
  pupil size will be monitored and recored using an infrared pupilometry system consisting of a camera, infrared lignt source, video monitor and video processing software, capturing pupil diameter as a real-time analogue signal (rate of 25 Hz). The pupil size variability will be used to estimate pain
change from baseline in heart rate during noxious stimulation | baseline and 5 minutes
  heart rate will be recorded before induction of anesthesia, just before nociceptive stimulation, then every 30 seconds up to the end of the five minutes after nociceptive stimulation. The heart rate measurement will be used to estimate pain.
Change from baseline in BIS (Bispectral Index) during noxious stimulation | baseline and 5 minutes
  bispectral index will be recorded before induction of anesthesia, just before nociceptive stimulation, then every 30 seconds up to the end of the five minutes after nociceptive stimulation. BIS will be used to estimate pain
change from baseline in systolic blood pressure during noxious baseline | baseline and 5 minutes
  Systolic blood pressure will be recorded before induction of anesthesia, just before nociceptive stimulation, then every 30 seconds up to the end of the five minutes after nociceptive stimulation. Systolic blood pressure measurement will be used to estimate pain
Change from baseline in diastolic blood pressure during noxious stimulation | basline and 5 minutes
  diastolic blood pressure will be recorded before induction of anesthesia, just before nociceptive stimulation, then every 30 seconds up to the end of the five minutes after nociceptive stimulation. diastolic blood pressure will be used to estimate pain

CONTACTS AND LOCATIONS:
Overall Officials: David Charier, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France